CLINICAL TRIAL: NCT05647967
Title: Evaluation of Regional Perfusion of Lung Consolidation Upon Lung Ultrasonography
Brief Title: Features of Regional Perfusion of Lung Consolidation
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Peking Union Medical College Hospital (Other)
Responsible Party: Sponsor
Other Study IDs: I-22PJ140
Record Dates: First submitted 2022-11-29; First posted 2022-12-13 (Actual); Last update posted 2022-12-13 (Actual); Status verified 2022-11

CONDITIONS: Lung Injury, Acute; Ultrasound Therapy; Complications
Keywords: lung consolidation, respiratory failure, perfusion
MeSH Terms: conditions — Acute Lung Injury; Respiratory Insufficiency | interventions — Ultrasonography

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- the consolidation perfusion/the consolidation size: Patients with respiratory failure and lung consolidation proved by chest imaging underwent lung ultrasound to evaluate the regional perfusion and the size of consolidation.
  Interventions: Diagnostic Test: Ultrasound

INTERVENTIONS:
Diagnostic Test: Ultrasound — Each patient underwent ultrasound after admission of ICU.

SUMMARY:
The aim of this study is to evaluate the potential usefulness of lung ultrasound to assess the size and perfusion of consolidation and explore their relationships with clinical outcome.

DETAILED DESCRIPTION:
Lung consolidation is one of the most causes of hypoxia in intensive care unit(ICU) settings. A quantitative measurement of consolidation would be extremely benefit for the clinical management in hypoxemia, both as an index of severity and to predict outcomes.In order to quantify the lung consolidation and its effect on clinical outcomes, a simple and quantitative scoring system of the size and perfusion of lung consolidation was proposed by lung ultrasound. Subjects with respiratory failure and lung consolidation proved by chest imaging underwent lung ultrasound examination. The size of consolidation and the richness of blood flow was computed upon lung ultrasound. The sensitivity, specificity and accuracy of the scoring system were calculated and compared to evaluate the diagnostic efficacy.

ELIGIBILITY:
Inclusion criteria:

1. Admission to ICU( 18yr<age<90yr);
2. Patients presented with acute respiratory failure;
3. Pulmonary consolidation by chest imaging (lung ultrasound, X ray or CT scan).

Exclusion criteria:

1. Hemodynamic instability (i.e., severe hypotension with systolic arterial pressure<60mmHg despite fluid expansion and vasoactive support; systolic arterial pressure>180mmHg; uncontrolled cardiac arrhythmias);
2. Severe thoracic trauma;
3. Coronavirus disease 2019;
4. Pulmonary artery hypertension and pregnancy.

Ages: 18 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: The study population consisted of adult(>18yr) patients admitted to the ICU. Patients presented with acute respiratory failure and pulmonary consolidation by chest imaging (lung ultrasound, X ray or CT scan) were eligible for inclusion. Acute respiratory failure was defined by at least one of the following criteria: PaO2/FiO2<300mmHg, breathing frequencies>30 breath/min, and could involve many potential causes of hypoxemia (e.g., sepsis, atelectasis, pneumonia, acute exacerbation of chronic lung disease).
Sampling Method: Non-Probability Sample
Enrollment: 200 (Estimated)
Dates: Start 2022-01-01 (Actual); Primary Completion 2023-12-31 (Estimated); Study Completion 2024-01-31 (Estimated)

PRIMARY OUTCOMES:
consolidation area index | through study completion, an average of 2 year
  The volume of consolidation was measured by consolidation area index (CAI) which is calculated from two-dimensional measures, namely the product of the core distance (from the bottom to the top of the screen) and the longitudinal distance (from the left to the right of the screen).
blood flow score | through study completion, an average of 2 year
  A semi-quantified scoring system based on the richness of flow signals was established. It identifies four progressive steps of blood signals, each corresponding to a score: no pulsatile blood flow-score 0; sparse dot-like blood flow-score 1; pronounced curvilinear vascularity-score 2; tree-like vascularity-score 3.

CONTACTS AND LOCATIONS:
Overall Officials: Huaiwu He, MD, Principal Investigator — Peking Union Medical College Hospital
Locations (1):
- Peking union medical college hospital, Beijing, Beijing Municipality, China

REFERENCES:
- [Derived] Wang N, Chi Y, Wang Q, Long Y, Liu D, Zhao Z, He H. Relationship between lung consolidation size measured by ultrasound and outcome in ICU patients with respiratory failure. BMC Pulm Med. 2025 Feb 26;25(1):91. doi: 10.1186/s12890-025-03564-6. PMID 40011857